CLINICAL TRIAL: NCT05685329
Title: An In Depth Study Examining Patterns in the Clinical Trial Experiences of Parkinson's Disease Patients
Brief Title: Determining Patterns In Trial Experiences of Parkinson's Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 87526739
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Parkinson's
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical studies is highly skewed towards particular demographic groups of people.

This study will invite several participants to gather a wide range of information on clinical trial experiences for Parkinson's Disease patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of Parkinson's Disease.

The data collected from this study will help improve future outcomes for all Parkinson's Disease patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient plans to participate in an interventional clinical trial for the condition of Parkinson's Disease
* Patient has been diagnosed with a type of Parkinson's Disease
* Patient is at least 50 to 80 years of age
* Patient has access to a home internet connection in order to provide regular updates through the course of the study

Exclusion Criteria:

* Patient has an ECOG score of 4 or higher
* Patient is not able to provide consistent digital updates as per study requirements
* Patient does not complete or agree to terms outlined in the Informed Consent Form

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an Parkinson's Disease clinical trial | 3 months
Rate of patients who remain in Parkinson's Disease clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reich SG, Savitt JM. Parkinson's Disease. Med Clin North Am. 2019 Mar;103(2):337-350. doi: 10.1016/j.mcna.2018.10.014. Epub 2018 Dec 3. PMID 30704685
- [Background] Armstrong MJ, Okun MS. Diagnosis and Treatment of Parkinson Disease: A Review. JAMA. 2020 Feb 11;323(6):548-560. doi: 10.1001/jama.2019.22360. PMID 32044947
- [Background] McFarthing K, Rafaloff G, Baptista M, Mursaleen L, Fuest R, Wyse RK, Stott SRW. Parkinson's Disease Drug Therapies in the Clinical Trial Pipeline: 2022 Update. J Parkinsons Dis. 2022;12(4):1073-1082. doi: 10.3233/JPD-229002. PMID 35527571

DOCUMENTS (1):
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT05685329/ICF_000.pdf